CLINICAL TRIAL: NCT03942094
Title: Efficacy and Safety of Nilotinib as the First-line Treatment for Patients With Newly Diagnosed Chronic-phase Chronic Myeloid Leukemia: a Prospective Study
Brief Title: Nilotinib for First-line Newly Diagnosed CML-CP Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Collaborators: Zhongshan People's Hospital, Guangdong, China (Other); Affiliated Hospital of Guangdong Medical University (Other); Huazhong University of Science and Technology Union Shenzhen Hospital (Unknown); Dongguan People's Hospital (Other Government); Longgang District People's Hospital of Shenzhen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nilotinib20190426
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Chronic Myeloid Leukemia, Chronic Phase; Nilotinib
Keywords: Nilotinib
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nilotinib (Experimental)
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — Nilotinib (Tasigna ®), capsules of 150 mg
  Nilotinib 2 capsules of 150 mg, orally, twice daily

SUMMARY:
This is a phase IIIb, multi-centre, single-arm, open-label, prospective study investigating the efficacy and safety of nilotinib as the first-line treatment for the adult patients with newly diagnosed chronic-phase chronic myeloid leukemia (CML-CP) in China. Nilotinib 300 mg BID will be provided in this study. The assessment for the primary efficacy endpoint will be performed at 18 months and the rate of patients obtaining MR4.5 will be measured at this time point. Secondary endpoints include the complete hematologic response(CHR) and the rates of major molecular reactions (MMR) by 3, 6, 9,12,18 and 24 months; event free survival (EFS); overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Newly diagnosed CP-CML within 6 months prior to study entry, positive Philadelphia chromosome or positive BCR-ABL (M-bcr transcript)
* Age ≥ 18 years old (no upper age limit given)
* CML-CP defined by primordial cells in peripheral blood or bone marrow <20%, basophils in peripheral blood <20%, platelets ≥100 x 109/L(≥100,000/mm3), except for hepatosplenomegaly
* Patient for whom treatment with Imatinib within 2 weeks is expected No other CML treatment except for hydroxyurea and/or anagrelide and/or IFN ECOG score 0 to 2
* Organ function defined by total serum bilirubin levels < 1.5 × the upper limit of the normal range (ULN), SGOT and SGPT < 2.5 UNL, creatinine < 1.5 × ULN, amylase and lipase ≤ 1.5 × ULN and alkaline phosphatase ≤ 2.5 × ULN not directly related to the CML
* Laboratory values defined by potassium ≥ LLN, magnesium ≥ LLN, phosphate ≥ LLN, total calcium (correction for serum albumin) ≥ LLN
* No planned allogeneic stem cell transplantation
* Signed informed consent

Exclusion Criteria:

* Patients confirmed to have a T315I mutation
* TKIs are not allowed to be treated prior to entering the study, unless the patient has an emergency pending the start of the study, and any dose of commercial imatinib may be used to the patient, but no more than 2 weeks
* Treatment with IFN for more than 3 mouths
* Impaired cardiac function including any of the following:

  1. Complete left bundle branch block
  2. Right bundle branch block plus left anterior hemiblock,bifascicular block
  3. Use of a ventricular-paced pacemaker
  4. Congenital long QT syndrome
  5. Clinically significant ventricular or atrial tachyarrhythmias
  6. Clinically significant resting bradycardia (<50 beats per minute)
  7. QTcF >450 msec on screening ECG.If QTcF >450 msec and electrolytes are not within normal ranges before nilotinib dosing, electrolytes should be corrected and then the patient rescreened for QTcF criterion
  8. Myocardial infarction within 12 months prior to starting nilotinib
  9. Other clinical significant heart disease (e.g. unstable angina,congestive heart failure,uncontrolled hypertension)
* Patients who are confirmed CNS infiltration by cytopathology
* Concurrent uncontrolled medical conditions (e.g. uncontrolled diabetes, active or uncontrolled infections)
* Congenital or acquired bleeding tendency
* Patients who have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Received other study medications within 30 days (defined as drugs that cannot be used based on approved indications)
* Patients unwilling or unable to comply with the protocol
* Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention
* Concomitant medications known to be strong inducers or inhibitors of the CYP450 Isoenzyme CYP3A4 (for example, erythromycin, ketoconazole, itraconazole, voriconazole, clarithromycin, telithromycin, ritonavir, and midazolam)
* Impaired gastrointestinal function or disease that may alter the absorption of study drug (e.g.ulcerative disease,uncontrolled nausea,vomiting and diarrhea,malabsorption syndrome,small bowel resection or gastric by-pass surgery)
* History of acute pancreatitis within 12 months or chronic pancreatitis
* History of acute or chronic diseases of Liver, pancreas or kidney
* Concomitant medications with potential QT prolongation
* Patients who are pregnant or breast feeding or women of reproductive potential not employing an effective method of birth control.Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to administration of nilotinib.Post menopausal women must be amenorrheic for at least 12 months in order to be considered of non-childbearing potential.Female patients must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Molecular response (MR) 4.5 at 18 months of nilotinib 300 mg twice a day | 18 months

SECONDARY OUTCOMES:
Molecular Response 4.5 at 3, 6, 9, 12, 24 months of nilotinib | 24 months
Major Molecular Response at 3, 6, 9, 12, 24 months of nilotinib | 24 months
Rate of CCyR (complete cytogenetic responses: bone marrow Philadelphie positive at 0 % on at least 20 metaphases) at 3, 6, 9, 12, 24 months of nilotinib. | 24 months
Event-free survival | 24 months
  Survival since randomization without any event defined as loss of CHR, loss of PCyR or CCyR, death from any cause, progression towards accelerated phase or blast crisis.
Overall survival | 24 months
  Survival without death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No